CLINICAL TRIAL: NCT01121198
Title: ASP1941 Phase I Study -Placebo-controlled, Single-dose and Repeated-dose Oral Administration Study in Healthy Adult Male Subjects-
Brief Title: A Study to Assess Safety and Tolerability of ASP1941 After Single and Repeated Administration in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Director, Astellas Pharma, Inc
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 1941-CL-0101
Record Dates: First submitted 2010-05-10; First posted 2010-05-12 (Estimated); Last update posted 2010-05-12 (Estimated); Status verified 2010-05

CONDITIONS: Healthy Volunteer; Pharmacokinetics of ASP1941
Keywords: Food effect
MeSH Terms: interventions — ipragliflozin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- ASP1941 single arm (Experimental)
  Interventions: Drug: ASP1941
- ASP1941 repeated arm (Experimental)
  Interventions: Drug: ASP1941
- placebo single arm (Placebo Comparator)
  Interventions: Drug: placebo
- placebo repeated arm (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: ASP1941 — oral
  Arms: ASP1941 repeated arm; ASP1941 single arm
Drug: placebo — oral
  Arms: placebo repeated arm; placebo single arm

SUMMARY:
This study is to assess the safety, tolerability, pharmacokinetics and pharmacodynamics of ASP1941 in healthy adult male subjects.

DETAILED DESCRIPTION:
This study consists of two parts. In part-1, a single oral dose of ASP1941 or placebo is administered to healthy adult male subjects to investigate the safety, tolerability, pharmacokinetics and pharmacodynamics in healthy adult males. In part-2, ASP1941 or placebo are is administered by a multiple dose regimen.

ELIGIBILITY:
Inclusion Criteria:

* Body weight: 50.0 kg ≤ weight < 85.0 kg
* Body mass index:17.6 ≤ BMI < 26.4
* Those who provided written informed consent themselves

Exclusion Criteria:

* Medical history of Hepatic disease, heart disease, respiratory disease, gastrointestinal disease, renal disease, cerebrovascular disease, malignant tumor or drug allergy
* Those whose blood pressure, pulse rate, body temperature or 12-lead ECG are in the abnormal range
* Those whose lab-test results are in the abnormal range
* Those who received medical treatment within 14 days prior to the study
* Those who attended another clinical study or a post-marketing clinical trial within 120 days before the study
* Those who have received ASP1941 before
* Those who have donated at least 400ml of whole blood within 90 days before the study, at least 200ml 30 days before the study or blood component within 14 days before the study
* Those within a fasting plasma glucose level of < 70mg/dL or 110 mg/dL or with an HbA1C. 5.8%

Ages: 20 Years to 44 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2006-12; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Safety assessed by adverse events, vital signs, 12-lead ECG and lab-tests | 72 hours after drug administration

SECONDARY OUTCOMES:
Plasma concentration of unchanged drug measured by blood sample | 72 hours after drug administration
Blood glucose level measured by blood sample | 72 hours after drug administration
Urinary glucose excretion level | 72 hours after drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Chair — Astellas Pharma Inc
Locations (1):
- Kantou, Japan